CLINICAL TRIAL: NCT04421248
Title: Anomalous Motor System Physiology in Attention Deficit Hyperactivity Disorder: Biomarker Validation and Modeling Domains of Function
Brief Title: Biomarker Validation in Motor System Physiology in Attention Deficit Hyperactivity Disorder
Acronym: AMPAIII
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Donald Gilbert, MD, MS, FAAN, FAAP (Other)
Collaborators: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor-Investigator, Donald Gilbert, MD, MS, FAAN, FAAP, Professor, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CHMC IRB 2020-0297
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Attention Deficit Hyperactivity Disorder Combined
MeSH Terms: interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: This is a randomized, blinded, placebo-controlled, single-dose crossover study. The objective is to estimate, in a rigorous, unbiased manner, the effect of 10 mg methylphenidate (MPH) on two putative biomarkers of ADHD, measured using Transcranial Magnetic Stimulation (TMS). Outcomes will be evaluated via repeated measures, mixed model analysis with MEP amplitude as the dependent variable and Treatment and Treatment-Sequence as class variables. Participants will include 144 children with ADHD. Study measures will also be compared in 70 matched, typically developing children who do not have ADHD and who will not receive methylphenidate or placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Preparation of identical single dose capsules of methylphenidate and placebo prepared by study pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Attention Deficit Hyperactivity Disorder (ADHD) (Experimental): 8 to 12 year old children diagnosed with ADHD. Randomized, blinded, single dose, placebo controlled, crossover trial.
  Interventions: Drug: Methylphenidate; Drug: Placebo
- Typically developing controls (TDC) (No Intervention): Typically developing controls - 8 to 12 year old children

INTERVENTIONS:
Drug: Methylphenidate — In ADHD participants only: blinded, randomized, placebo-controlled single dose, crossover on separate days separated by at least one week.
  Other Names: Ritalin
  Arms: Attention Deficit Hyperactivity Disorder (ADHD)
Drug: Placebo — In ADHD participants only: blinded, randomized, placebo-controlled, single dose, crossover on separate days separated by at least one week.
  Arms: Attention Deficit Hyperactivity Disorder (ADHD)

SUMMARY:
Attention-Deficit/Hyperactivity Disorder (ADHD) is the most commonly diagnosed neurobehavioral disorder in childhood. Children with ADHD struggle in school due to problems with attention and high levels of impulsivity and hyperactivity. They are at substantially increased risk for long-term difficulties into adulthood, including academic underachievement, substance abuse, and criminal behavior. The diagnosis of ADHD, which is based on subjective ratings by parents and teachers, likely results from multiple different, overlapping differences in circuits of the brain responsible for attention and impulse control. However, we do not have any scientific or clinical tests that allow us to understand these circuits. In an effort to improve ADHD outcomes, we have used a technology called Transcranial Magnetic Stimulation (TMS) to identify highly reliable measurements of brain function. We have identified two very promising measures that are abnormal in children with ADHD and, importantly, also predict the severity of ADHD behaviors. The goal of this project is to determine if these two TMS measurements could be used to help better guide ADHD treatment. To do this, we will perform three investigations in 8 to 12 year old children to determine: 1) test-retest reliability; 2) pharmacologic responsiveness; and 3) correlations with two domains of function relevant to ADHD: "Cognitive Control" and "Emotional Valence." Through these investigations, we aim to determine whether these two TMS brain measures are reliable and meaningful enough to be used to help improve precision of individually-targeted and effective ADHD treatments.

DETAILED DESCRIPTION:
4.2. NARRATIVE STUDY DESCRIPTION

Summary This is a randomized, blinded, placebo-controlled, single-dose crossover study. The objective is to estimate, in a rigorous, unbiased manner, the effect of 10 mg methylphenidate (MPH) on two putative biomarkers of ADHD, measured using Transcranial Magnetic Stimulation (TMS). Two other aims of this larger study, quantifying test-retest reliability and linking TMS biomarkers to RDoC domains of cognitive control and emotional valence, are not directly part of the clinical trial and are fully described in the research strategy.

Doctors use observations and subjective rating scales both to diagnose Attention Deficit Hyperactivity Disorder (ADHD) and to make decisions about medical or behavioral treatments. This study addresses the possibility that in children with ADHD, brain-based measurements, or biomarkers, could be useful for diagnosis and treatment decisions. These biomarkers are Short Interval Cortical Inhibition (SICI) and Task-Related Up-Modulation (TRUM). These biomarkers may allow clinicians to identify that a child has a "type" of ADHD which might respond more effectively to treatments that are precisely and individually targeted. Thus it is important to estimate the effects of commonly prescribed treatments on SICI and TRUM. This protocol aims to determine the effects of a single 10 mg dose of MPH, a stimulant medication widely prescribed to treat ADHD, on SICI and TRUM.

Assignment of participants For each child with ADHD, participation in the study will consist of three visits. Treatment occurs as a single dose on visits 2 and 3. All participants will receive both placebo and 10 mg MPH. Order will be counterbalanced.

Population Sample At the two study sites, Cincinnati Children's Hospital Medical Center (CCHMC) and the Kennedy Krieger Institute (KKI), we will recruit 144 pre-pubescent children, ages 8 years 0 months to 12 years 11 months, with ADHD. We estimate a total of 120 participants will participate in the full study. All recruitment methods will conform to CCHMC Institutional Review Board (IRB) and HIPAA requirements. The study will be approved by the CCHMC Institutional IRB. Children with ADHD will be primarily recruited through community resources, including local chapters of the Children with ADHD (CHADD), local public and private schools, as well as multiple clinics at CCHMC and KKI.

Study Flow During the first study visit, participants will provide informed consent. They will then complete diagnostic and psychoeducational testing. The parent/guardian will complete standardized questionnaires and a comprehensive psychiatric diagnostic interview with a trained and research reliable psychology associate under the supervision of a neuropsychologist at each site.

At visit 1: if determined to be eligible to continue, visits 2 and 3 will be scheduled at 2-week intervals.

At visit 2: participant will undergo pre-dose TMS for measures of SICI and TRUM, receive either MPH or placebo, then undergo post-dose TMS.

At visit 3: participant will undergo pre-dose TMS measures of SICI and TRUM (test/re-test assessment), receive the opposite treatment of either MPH or placebo, then undergo post-dose TMS.

Intervention - MPH versus Placebo Procedures

The MPH and the placebo will be prepared by the study pharmacy at each site so that they appear identical. Neither the child, the parent, nor the investigators will know which treatment is given. The study pharmacy will randomize children into two groups, without disclosing this information to the researchers or participants. Group 1 will receive MPH on the first treatment visit (visit 2 of the study) and placebo the second. Group 2 will receive placebo on the first treatment visit and MPH the second.

Note: for comparison and validation of the study measures, 70 children who are typically developing and do not have ADHD will also be enrolled. These control participants will not receive methylphenidate or placebo, however.

ELIGIBILITY:
Inclusion Criteria:

* Either gender, any race, ethnicity or socioeconomic status
* Currently between 8 years 0 months and 12 years, 11 months, 30 days
* Willing to answer questions about ADHD and related diagnoses
* For children with ADHD prescribed stimulant medications, willing to suspend taking medications as specified in the study procedures
* For children with ADHD, willing to participate in the single dose, randomized crossover study to probe acute effects of methylphenidate on biomarkers
* Right hand dominant (predominately right-handed)
* Able to participate in and sign an informed consent
* ADHD inclusion: The diagnosis of ADHD will be based on Diagnostic and Statistical Manual version 5 (DSM-5) criteria using standard rating scales and a structured diagnostic interview. Oppositional Defiant Disorder is permitted; Conduct disorder is excluded.
* Typically Developing (healthy control) inclusion: Free of ADHD or other developmental or psychiatric disorders based on DSM-5 criteria using standard rating scales and a structured diagnostic interview.

Exclusion Criteria:

* Known diagnosis of mental retardation, cerebral palsy, Autism Spectrum Disorder, traumatic brain injury, brain tumor, epilepsy, or other serious neurological disorder.
* Major Depression, Bipolar Disorder, Conduct Disorder, Adjustment Disorder, other Anxiety Disorders, or other developmental psychiatric diagnoses.
* For females, onset of menses, pregnancy.
* Current use of antidepressants, non-stimulant ADHD medications, dopamine blocking agents, mood stabilizers.
* Implanted brain stimulator, vagal nerve stimulator, ventriculo-peritoneal shunt, cardiac pacemaker, or implanted medication port.
* Diagnosis of a speech/language disorder or a Reading Disability (RD).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 214 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Transcranial Magnetic Stimulation (TMS)-evoked Short Interval Cortical Inhibition (SICI) Test-Retest Reliability | less than one month
  A ratio of amplitudes of motor evoked potentials from paired (inhibitory) and single TMS pulses, obtained from dominant motor cortex with hand at rest
Transcranial Magnetic Stimulation (TMS)-evoked Task Related Up Modulation (TRUM) Test-Retest Reliability | less than one month
  A ratio of amplitudes of motor evoked potentials during engagement in a response inhibition task versus rest, obtained from dominant motor cortex

CONTACTS AND LOCATIONS:
Overall Officials: Donald L Gilbert, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Stewart H Mostofsky, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (2):
- United States (2):
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Sharing of individual participant data (IPD) will occur through the National Institute of Mental Health (NIMH) Data Archive, consistent with the NIMH Data Sharing Policy. This includes all raw and analyzed data, including clinical, phenotypic, and neurophysiological biomarker data, which will be de-identified and deposited in the NIMH Data Archive (NDA). Data from research subjects will include Required Data Elements: 1) NDA Global Unique Identifier assigned to participants (GUID); 2) the study's internal subject identifier (Src_subject_id); 3) interview age in months (interview_age); 4) data collection date (interview_date); and 5) birth sex.
Supporting Information: Study Protocol, SAP
Time Frame: Data uploads to the NIMH Data Archive from the study will occur every 6 months, consistent with the NIMH Data Sharing Policy.
Access Criteria: Determined by NIMH.

REFERENCES:
- [Background] Doherty AC, Huddleston DA, Horn PS, Ratner N, Simpson BN, Schorry EK, Aschbacher-Smith L, Prada CE, Gilbert DL. Motor Function and Physiology in Youth With Neurofibromatosis Type 1. Pediatr Neurol. 2023 Jun;143:34-43. doi: 10.1016/j.pediatrneurol.2023.02.014. Epub 2023 Mar 3. PMID 36996759
- [Background] Luo Y, Adamek JH, Crocetti D, Mostofsky SH, Ewen JB. Dissociation in Neural Correlates of Hyperactive/Impulsive vs. Inattentive Symptoms in Attention-Deficit/Hyperactivity Disorder. Front Neurosci. 2022 Jun 22;16:893239. doi: 10.3389/fnins.2022.893239. eCollection 2022. PMID 35812240
- [Background] Luo Y, Chen C, Adamek JH, Crocetti D, Mostofsky SH, Ewen JB. Altered cortical activation associated with mirror overflow driven by non-dominant hand movement in attention-deficit/hyperactivity disorder. Prog Neuropsychopharmacol Biol Psychiatry. 2022 Jan 10;112:110433. doi: 10.1016/j.pnpbp.2021.110433. Epub 2021 Aug 27. PMID 34454990
- [Background] Chen C, Rosch KS, Seymour KE, Crocetti D, Mahone EM, Mostofsky SH. Sex Effects on Mirror Overflow during Finger Tapping in Children with ADHD. J Int Neuropsychol Soc. 2022 Apr;28(4):371-381. doi: 10.1017/S1355617721000576. Epub 2021 May 17. PMID 33998435
- [Background] Nikolaidis A, He X, Pekar J, Rosch K, Mostofsky SH. Frontal corticostriatal functional connectivity reveals task positive and negative network dysregulation in relation to ADHD, sex, and inhibitory control. Dev Cogn Neurosci. 2022 Apr;54:101101. doi: 10.1016/j.dcn.2022.101101. Epub 2022 Mar 23. PMID 35338900
- [Background] Thapaliya G, Carnell S, Mostofsky SH, Rosch KS. Neurobehavioral phenotypes of delay discounting and cognitive control in child attention-deficit/hyperactivity disorder and obesity: Shared or distinct? Pediatr Obes. 2023 Apr;18(4):e13001. doi: 10.1111/ijpo.13001. Epub 2023 Jan 18. PMID 36655309